CLINICAL TRIAL: NCT05027672
Title: Randomised Phase II Study to Assess the Immunogenicity and Safety of Heterologous SARS-CoV-2 Vaccine Schedules (rAd26-rAd5, rAd26-rAd26, rAd26-ChAdOx1 and rAd26-mRNA-1273).
Brief Title: Strategies for Combining the First Component of Sputnik V With Other Adenoviral or mRNA-based Vaccines.
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Ministerio de Salud de Ciudad Autónoma de Buenos Aires (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 5143_3
Record Dates: First submitted 2021-08-18; First posted 2021-08-30 (Actual); Last update posted 2021-08-30 (Actual); Status verified 2021-08

CONDITIONS: COVID-19 Vaccines
Keywords: COVID-19 Serological Testing
MeSH Terms: interventions — Gam-COVID-Vac vaccine; ChAdOx1 nCoV-19

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: All personnel involved in antibody determination shall remain blinded to the assigned strategy.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Gam-COVID-Vac (rAd26) / Gam-COVID-Vac (rAd5) (Active Comparator): At the time of randomisation, patients in this arm receive a second dose of Sputnik V (rAd5) vaccine component two.
  Interventions: Drug: Gam-COVID-Vac (rAd26) / Gam-COVID-Vac (rAd5)
- Gam-COVID-Vac / ChAdOx1 nCoV-19 (Experimental): At the time of randomisation, patients in this arm receive Astra Zeneca's vaccine (ChAdOx1 nCoV-19) as a second dose.
  Interventions: Drug: Gam-COVID-Vac (rAd26) / Gam-COVID-Vac (rAd5)
- Gam-COVID-Vac / Gam-COVID-Vac (rAd26) (Experimental): At the time of randomisation, patients in this arm receive a second dose of a repeat of the first component of the Sputnik V vaccine (rAd26) as a second dose.
  Interventions: Drug: Gam-COVID-Vac (rAd26) / Gam-COVID-Vac (rAd5)
- Gam-COVID-Vac / mARN-1273 (Experimental): At the time of randomisation, patients in this arm receive as a second dose the vaccine produced by Moderna (mRNA-1273).
  Interventions: Drug: Gam-COVID-Vac (rAd26) / Gam-COVID-Vac (rAd5)

INTERVENTIONS:
Drug: Gam-COVID-Vac (rAd26) / Gam-COVID-Vac (rAd5) — A comparison of antibody levels against protein S will be performed using the Gam-COVID-Vac / Gam-COVID-Vac group as a control group and all other interventions as comparators.Comparisons will be made by contrasting the geometric means of antibody levels between each of the study arms. In addition, comparisons will be made as to whether or not the median antibody values of the alternative treatment groups are lower than: a) the 25th percentile of the median antibody value of the Gam COVID combination and b) whether the lower limit of the confidence interval of the differences in the GMC rate is lower than the conventional cut-off point of non-inferiority set at 0.67.
  Other Names: Gam-COVID-Vac (rAd26) / ChAdOx1 nCoV-19; Gam-COVID-Vac (rAd26) / Gam-COVID-Vac (rAd26); Gam-COVID-Vac (rAd26) / mARN-1273

SUMMARY:
To determine whether a heterologous vaccination regimen in individuals with no known previous history of COVID-19 is non-inferior to that observed with counterpart regimens currently in use in Argentina among persons aged 21 to 65 years

DETAILED DESCRIPTION:
The Covid-19 disease caused by the SARS-COV 2 virus has caused a pandemic with more than 180 million cases worldwide and more than 4 million deaths. In Argentina, this pandemic has had a significant impact, with about 4.5 million cases and about 95,000 deaths. In no more than nine months, medical science developed different vaccines to prevent new cases and mitigate this pandemic.

At the time of the presentation of this research protocol, there are four vaccines for the prevention of COVID-19 approved for emergency use by the National Administration of Medicines, Food and Medical Technology (ANMAT). Argentina recently received a donation of 3.2 million doses of Moderna (mRNA-1273) vaccine from the US government. This vaccine was approved for emergency use in the context of the pandemic. All require the administration of two doses with an administration interval of at least 21 days.

All these vaccines were designed to be used with a homologous two-dose regimen. However, for both logistical and biomedical reasons, the need to use vaccines in heterologous regimens (one dose of one vaccine and a second dose of another vaccine) is emerging worldwide. The efficacy and safety of this type of regimen has not yet been demonstrated.

In Argentina, there are a large number of people who currently have one dose of Gam-COVID-Vac vaccine and who - even after a period of ≥21 days - have not received the second component. At the same time, the provision of the second component of the Gam-COVID-Vac vaccine is delayed due to production and distribution logistics.

As of 08/02/2021, among the universe of people vaccinated with Gam-COVID, residents of CABA, vaccinated in establishments in the City of Buenos Aires - and excluding deceased and infected people - there were a total of 332,291 people with one dose and ≥22 days since the first dose was administered. In a context of high viral circulation, it is desirable to try to vaccinate as much of the population as possible with a full schedule in the shortest possible time. In addition, new variants of SARS-COV2 virus possessing the E384K genomic variant such as the gamma strain (formerly Manaus), the beta strain (known as South African) and the Delta strain (also known as Indian) have the ability to evade the immune system and therefore most laboratories that have developed vaccines recognise that the efficacy of the vaccines requires two doses.

This study will attempt to determine whether administration of a heterologous regimen combining a first dose of Gam-COVID-Vac the repetition of the first component of the Gam-COVID-Vac vaccine (rAd26) or the administration of an RNA vaccine (mRNA-1273) resulted in a non inferiority result that the classic and recomended protocol based on two dosis of Gam-COVID-Vac (rAd26-rAd5) .

The present protocol is therefore oriented to respond to a practical management need and to guarantee the best possible protection to the population through two doses, which is what is considered worldwide as "complete vaccination" according to WHO for the vaccines used by Argentina. The proposed protocol is a pragmatic and public health oriented clinical trial, whose primary objective is to establish whether there are indicators that allow the implementation of a heterologous vaccination scheme. For this, a surrogate endpoint will be used, which is immunogenicity measured by the presence of antibodies against protein S. In addition, the safety of the combination will be evaluated in terms of monitoring self-reported and non-self-reported clinical events by patients.

ELIGIBILITY:
Inclusion Criteria:

* Persons who have received a dose of Gam-COVID-Vac more than 30 days and:
* Age > 21 and <66 years.
* Both genders.
* Who have voluntarily agreed to participate in the clinical trial and have provided informed consent.

Exclusion Criteria:

* Known history of COVID in the 6 months prior to study inclusion.
* Known or suspected immunocompromised status by the study investigator for any cause.
* Use of oral or parenteral corticosteroids in the last 30 days.
* Known history of allergy to any vaccine.
* History of anaphylaxis.
* Pregnant or lactating women.
* Known history of autoimmune diseases.
* Persons under treatment for any neoplastic disease within the last 6 months.
* Any serious illness or condition at the discretion of the study investigator (including but not limited to the presence of chronic obstructive pulmonary disease, heart failure, poorly controlled hypertension, poorly controlled diabetes, renal failure).
* Planned medical procedures within two months of randomisation.
* Previous vaccination within the last 30 days with any vaccine.
* Known participation in an ongoing clinical trial.
* Ongoing acute illness.
* Fever (≥37.8 C) at the time of randomisation.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 348 (Actual)
Dates: Start 2021-07-30 (Actual); Primary Completion 2021-08-30 (Estimated); Study Completion 2021-09-06 (Estimated)

PRIMARY OUTCOMES:
ELISA assessment of concentration of IgG anti Spike (UI/ml) at 28 days. | 28 days
  To determine whether a heterologous vaccination regimen in individuals with no known previous history of COVID-19 is non-inferior to that observed with currently used counterpart regimens.
  The assessment of the antibody concentration in each of the study arms will be measured by measuring the IgG antibody concentration using ELISA expressed in IU/ml. Additionally, geometric mean concentration ratio will be measured comparing the ratio between Sputnik vaccination and that obtained in each study arm.
Serious adverse events Adverse events of special interest | 28 days
  To report the combine and specific rate of serious adverse defined as death for any reason, any life-threatening event or any event that require inpatient hospitalization.

SECONDARY OUTCOMES:
Neutralising antibodies against SARS-CoV-2 | 28 days
  Neutralising antibody titres at baseline, 14 days and 28 days after randomisation will be measured in all participants.

CONTACTS AND LOCATIONS:
Locations (2):
- Argentina (2):
  - Ministerio de Salud de la Ciudad Autónoma de Buenos Aires, Buenos Aires, CBA
  - Ministerio de Salud de la Ciudad Autónoma de Buenos Aires, Buenos Aires

IPD SHARING:
Plan to Share IPD: No